CLINICAL TRIAL: NCT02708251
Title: Topical Glyceryl Trinitrate Versus Lidocaine Cream as Analgesia for IUD Insertion: A Randomized Controlled Trial
Brief Title: Glyceryl Trinitrate Versus Lidocaine Cream for IUD Insertion
Acronym: GTN-IUD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GTN
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: IUD Insertion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- glyceryl trinitrate cream (Experimental): The clinician will perform a bimanual examination, place the speculum, and cleanse the cervix with Betadine. 1 mL glyceryl trinitrate cream will be placed on the cervix at the anterior lip and 1 mL in the cervix up to the level of the internal os using cotton swab.
  Interventions: Drug: glyceryl trinitrate cream
- lidocaine cream (Experimental): The clinician will perform a bimanual examination, place the speculum, and cleanse the cervix with Betadine. 1 mL lidocaine creamwill be placed on the cervix at the anterior lip and 1 mL in the cervix up to the level of the internal os using cotton swab.
  Interventions: Drug: lidocaine cream
- placebo cream (Placebo Comparator): The clinician will perform a bimanual examination, place the speculum, and cleanse the cervix with Betadine.1 mL placebo cream will be placed on the cervix at the anterior lip and 1 mL in the cervix up to the level of the internal os using cotton swab.
  Interventions: Drug: placebo cream

INTERVENTIONS:
Drug: glyceryl trinitrate cream
  Arms: glyceryl trinitrate cream
Drug: lidocaine cream
  Arms: lidocaine cream
Drug: placebo cream
  Arms: placebo cream

SUMMARY:
The intrauterine device (IUD) is a long-acting, highly effective, reversible contraceptive method that may be underutilized due to fear of pain during insertion. Although providers frequently prescribe non-steroidal anti-inflammatory drugs (NSAIDs) for IUD insertion, there is no evidence for any pain reduction. Women can experience high levels of pain when the IUD is placed inside the uterus, and fear of this pain could be a reason that women decide not to use this method.

ELIGIBILITY:
Inclusion criteria:

1. Women not taken analgesics or anxiolytics in the 24 hours prior insertion
2. Women not taken misoprostol prior to IUD insertion
3. No contraindication to or history of allergic reaction to lidocaine or NO donors.
4. Women who will accept to participate in the study

Exclusion criteria:

1. Lidocaine allergy
2. History of migraine or chronic headache
3. Any contraindication to IUD placement

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Mean pain score during IUD insertion | 3 minutes

SECONDARY OUTCOMES:
Patient satisfaction score after the procedure | 3 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Abbas AM, Ragab E, Abd Ellah NH, Sabra A, Ali SS, Mohamed A, Yosef AH. Effect of topical glyceryl trinitrate cream on pain perception during intrauterine device insertion in multiparous women: A randomized double-blinded placebo-controlled study. J Gynecol Obstet Hum Reprod. 2019 Nov;48(9):715-718. doi: 10.1016/j.jogoh.2019.03.007. Epub 2019 Mar 18. PMID 30898632